CLINICAL TRIAL: NCT06282185
Title: SUPERvised Three-month Exercise Program in MEN With Prostate cAncer Receiving Androgen-deprivaTioN thERapy
Acronym: Superman
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: no recruitments
Sponsor: Canisius-Wilhelmina Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CanisiusWH
Record Dates: First submitted 2023-01-16; First posted 2024-02-28 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Prostatic Neoplasms; Metastasis
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: randomized controlled trial with an intervention arm and an usual care group
Who Masked: Investigator, Outcomes Assessor
Masking Description: In a single blinded (investigators blinded to group allocation) randomized controlled pilot, conducted in the CWZ, 20 patients with advanced prostate cancer will be randomized across: 1) supervised training program for twelve weeks + usual care + advice about exercise, or 2) usual care + advice about exercise.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention (Experimental): supervised training program for twelve weeks + usual care + advice about exercise
  Interventions: Other: Physiotherapy
- usual care (No Intervention): usual care + advice about exercise

INTERVENTIONS:
Other: Physiotherapy — supervised training program for twelve weeks + usual care + advice about exercise
  Arms: intervention

SUMMARY:
The goal of this single blind placebo-controlled intervention study is to examine the impact of a supervised training program on disease-related quality of life and physical fitness in patient with advanced prostate cancer compared to usual care. The main question[s] it aims to answer are:

* What is the impact of exercise on quality of life
* What is the impact of exercise on physical fitness

Participants will have an individual training program with supervised training by physiotherapists.

Researchers will compare with usual care to see if advice about exercise has significant less effect than an supervised training program.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Age > 18 years old
* Able to read and complete questionnaires in Dutch
* Proven histologically and /or radiologically metastatic prostate cancer (TxNxM1)

Exclusion Criteria:

* Other cancers
* Clinicians' judgement
* Age >80 years old or not able to walk 400m
* Structural exercise (moderate-intensity exercise more than 150 minutes a week) during the past 3 months
* Musculoskeletal, cardiovascular, or neurological disorders that could inhibit them from exercising
* Spinal cord compression, history of pathological fractures

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
change of quality of life assessed with EPIC26 (0-100 points) | 6 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaire is used: Expanded Prostate Cancer Index Composite (EPIC26). With higher scores representing better disease-related quality of life.
change of quality of life assessed with EPIC26 (0-100 points) | 3 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaire is used: Expanded Prostate Cancer Index Composite (EPIC26). With higher scores representing better disease-related quality of life.
change of quality of life assessed with EORTC QLQ-C30 (0-100 points per scale) | 6 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaires are used: European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC QLQ-C30). A higher score represents a higher response level. So a higher score for the functional scale represents a higher level of physical functioning but a higher score for the symptoms scale represents a higher level of symptoms.
change of quality of life assessed with EORTC QLQ-C30 (0-100 points per scale) | 3 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaires are used: European Organization for Research and Treatment for Cancer Quality of Life Questionnaire (EORTC QLQ-C30). A higher score represents a higher response level. So a higher score for the functional scale represents a higher level of physical functioning but a higher score for the symptoms scale represents a higher level of symptoms.

SECONDARY OUTCOMES:
change of physical fitness in maximum uptake of oxygen in ml/kg/min | 6 months
  Assessment of the effectiveness of a supervised training program on cardiopulmonary fitness in patients with metastatic prostate cancer compared to usual care.
change of physical fitness in maximum uptake of oxygen in ml/kg/min | 3 months
  Assessment of the effectiveness of a supervised training program on cardiopulmonary fitness and body composition in patients with metastatic prostate cancer compared to usual care.
change of physical fitness in fat percentage | 3 months
  change in body composition in patients with metastatic prostate cancer compared to usual care.
change of physical fitness in fat percentage | 6 months
  change in body composition in patients with metastatic prostate cancer compared to usual care.
change of fitness assessed with IPAQ-sh (categories (1-3) and continues (MET-minutes)) | 3 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaires are used: Short Hebrew International Physical Activity Questionnaire (IPAQ-sh). Both categorical and continuous indicators of physical activity will be used from the IPAQ short form. There are three categories:1. inactive, 2. minimally active, 3. HEPA active (health enhancing physical activity; a high active category). The continuous score is reported in median MET-minutes (metabolic equivalent of task-minutes). For categorical and continuous score is a higher score equivalent of higher physical functioning.
change of fitness assessed with IPAQ-sh (categories (1-3) and continues (MET-minutes)) | 6 months
  To examine the impact of a supervised training program on disease-related quality of life in patient with advanced prostate cancer compared to usual care. The following questionnaires are used: Short Hebrew International Physical Activity Questionnaire (IPAQ-sh). Both categorical and continuous indicators of physical activity will be used from the IPAQ short form. There are three categories:1. inactive, 2. minimally active, 3. HEPA active (health enhancing physical activity; a high active category). The continuous score is reported in median MET-minutes (metabolic equivalent of task-minutes). For categorical and continuous score is a higher score equivalent of higher physical functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Paul van Basten, Dr. MD, Principal Investigator — Canisius Wilhelmina Ziekenhuis (CWZ)
Locations (1):
- Canisius Wilhelmina Ziekenhuis (CWZ), Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No